CLINICAL TRIAL: NCT03065335
Title: Neuropharmacologic Imaging and Biomarker Assessments of Response to Acute and Repeated-Dosed Ketamine Infusions in Major Depressive Disorder
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 170060; 17-M-0060
Record Dates: First submitted 2017-02-24; First posted 2017-02-27 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-10-24

CONDITIONS: Healthy Volunteer; Major Depressive Disorder; Depression
Keywords: Magnetic Resonance Imaging; Magnetoencephalography; Major Depressive Disorder; Ketamine; Neuropharmacology
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Ketamine; Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (8):
- Metabolites Substudy (Experimental): Open-label, single dose of 0.5 mg/kg IV ketamine
  Interventions: Drug: Ketamine
- Phase I (Experimental): Medication taper, drug-free period, and baseline assessments
  Interventions: Device: Cobot TS MV robotic arm for TMS
- Phase II, Arm 1 (Experimental): Double-blind, single dose of 0.5 mg/kg IV ketamine
  Interventions: Drug: Ketamine; Device: Cobot TS MV robotic arm for TMS
- Phase II, Arm 1b (Experimental): Double-blind, single dose of 0.5 mg/kg IV ketamine, concurrently with fMRI+EEG or MEG
  Interventions: Drug: Ketamine; Device: Cobot TS MV robotic arm for TMS
- Phase II, Arm 2 (Placebo Comparator): Double-blind, single dose of 0.5 mg/kg IV saline
  Interventions: Other: Placebo; Device: Cobot TS MV robotic arm for TMS
- Phase II, Arm 2b (Placebo Comparator): Double-blind, single dose of 0.5 mg/kg IV saline, concurrently with fMRI+EEG or MEG.
  Interventions: Other: Placebo; Device: Cobot TS MV robotic arm for TMS
- Phase III (Experimental): Double-blind, repeated dose of 0.5 mg/kg or 0.1 mg/kg IV ketamine
  Interventions: Drug: Ketamine; Device: NeurOptics PLRTM-30000 Pupillometer
- Phase IV (No Intervention): Follow-up evaluations

INTERVENTIONS:
Drug: Ketamine — N-methyl-D-aspartate (NMDA) glutamate receptor (NMDA-R) antagonist
  Arms: Metabolites Substudy; Phase II, Arm 1; Phase II, Arm 1b; Phase III
Other: Placebo — Placebo comparator
  Arms: Phase II, Arm 2; Phase II, Arm 2b
Device: Cobot TS MV robotic arm for TMS — TMS-Cobot TS MV [Axilum Robotics] robotic arm for spatial positioning and orientation of the TMS coil
  Arms: Phase I; Phase II, Arm 1; Phase II, Arm 1b; Phase II, Arm 2; Phase II, Arm 2b
Device: NeurOptics PLRTM-30000 Pupillometer — The Neu-rOptics PLRTM-3000 Pupillometer will use quantitative infrared technology to objectively and accurately measure pupil size and dynamics.
  Arms: Phase III

SUMMARY:
Background:

Most medications that treat depression take weeks or months to work. Researchers want to develop fast-acting treatments. One dose of ketamine has a rapid antidepressant effect. For most people, this lasts a week or less. Repeated doses of ketamine may help maintain this effect.

Objective:

Main Study: To study the effects of ketamine in treating depression.

Ketamine Metabolites Substudy: To study how ketamine effects brain chemistry.

To study how ketamine effects the brain. This is done by looking at metabolites, which are created when a drug is broken down.

Eligibility:

Main Study: People ages 18-65 with major depressive disorder and healthy volunteers

Ketamine Metabolites Substudy: Healthy volunteers ages 18-65

Design:

Main Study:

Participants will be screened in another study, with:

* Medical and psychiatric history
* Psychiatric and physical exam
* Blood, urine, and heart tests

Participants will be inpatients at NIH for 4 phases totaling 14-20 weeks.

Phase I (2-7 weeks):

* Gradually stop current medications
* MRI: Participants lie and perform tasks in a machine that takes pictures of the body.
* Mood and thinking tests
* Blood and urine tests
* Sleep test: Monitors on the skin record brain waves, breathing, heart rate, and movement during sleep.
* Transcranial magnetic stimulation: A coil on the scalp gives an electrical current that affects brain activity.
* Stress tests: Electrodes on the skin measure reactions to loud noises or electric shocks.

Phase I tests are repeated in Phases II and III and in the final visit.

Phase II (4-5 weeks):

* 4 weekly IV infusions of ketamine or a placebo during an MRI or MEG. For the MEG, a cone over the head records brain activity.

Phase III (optional):

* 8 infusions of ketamine over 4 weeks

Phase IV (optional):

* Symptoms monitoring for 4 weeks
* Participants will have a final visit. They will be offered standard treatment at NIH for up to 2 months.

Ketamine Metabolites Substudy:

Participants will be screened in another study, with:

* Medical and psychiatric history
* Psychiatric and physical exam
* Blood, urine, and heart tests

Participants will be inpatients at NIH for 4 days.

Study Procedures:

Mood and thinking tests

Blood and urine tests

1 infusion of ketamine

Spinal tap and spinal catheter: Used to get samples of cerebrospinal fluid (CSF). This is a fluid that moves around and within the brain and spinal cord. Studying CSF will help us learn how ketamine effects brain chemistry

DETAILED DESCRIPTION:
Objective

The current protocol has a two-fold purpose. In the pharmacodynamic imaging phase, we will investigate the neuropharmacodynamics of acute intravenous ketamine administration in patients with major depressive disorder (MDD) and healthy volunteers (HV) using functional MRI (fMRI) and electrophysiological modalities [electroencephalography (EEG) and magnetoencephalography (MEG)]. We will also investigate if specific signatures from functional neuroimaging, transcranial magnetic stimulation (TMS) associated evoked potentials (TMS-EP), sleep EEG (S-EEG), and psychophysiologic responses can be used to classify specific subpopulations of patients with MDD; preliminary findings from such an approach may be important in forging further studies identifying those who will respond to ketamine infusions. In the repeat-dosing phase, we will expand upon our previous findings of the immediate efficacy of glutamatergic modulators by investigating the safety and efficacy of repeated dose administrations of ketamine in MDD patients. We will include all MDD patients regardless of antidepressant response to single infusions of ketamine to allow for potential identification of patients who are able to attain and/or maintain a response over a series of infusions. To reduce any potential biases due to partial blinding, all patients will be randomized into groups to receive ketamine at either 0.5 mg/kg or 0.1 mg/kg (an active comparator).

Study Population

The study consists of 50 patients with treatment-resistant MDD between 18 and 65 years old and 50 age/gender matched HVs. Within the MDD group, 25 patients will be enrolled into each group in the repeat-dosing phase. An addition 50 HVs will participate in the Ketamine Metabolites Substudy.

Study Design

This study is a Phase I Clinical Trial that comprises four phases.

Phase I includes screening, medication taper (patients, as needed), medication-free period (patients), and baseline assessments, including optional TMS-EP, S-EEG, the None, Predictive, Unpredictive (NPU)-threat test, non-brain imaging cognitive tasks, and blood samples for plasma neurochemicals and peripheral blood biomarkers.

In Phase II, all subjects (patients with MDD and HVs) will receive an alternating series of placebo and ketamine infusions, once per week, for a total of 4 infusions (2 ketamine, 2 placebo). Concurrently with each infusion, subjects will be administered either resting-state fMRI with simultaneous EEG, or resting state MEG recording, thus each subject receives fMRI+EEG and MEG for both a placebo and ketamine infusion. Participants may also undergo optional sEEG, non-brain imaging cognitive tasks, TMS-EP, and NPU.

Phase III involves MDD patients whose depression symptoms relapsed after the final infusion in Phase II. Patients whose symptoms did not relapse may receive an additional one-week washout prior to participating in Phase III. Subjects will be randomized to receive ketamine at 0.5 or 0.1 mg/kg twice weekly for 4 weeks (total of 8 infusions). Participants may undergo optional fMRI, S-EEG, MEG, non-brain imaging cognitive tasks, TMS-EP, pupillometry, and NPU at time points between infusions. Clinical rating scales will assess depression symptomology and blood will be drawn for pharmacokinetics testing and biomarker analyses.

Phase IV includes patients who completed Phase III and who are responders. These patients will be followed up for an additional 4 weeks, or until relapse (whichever comes first), to determine durability of response. The final study day will include rating scales, medical evaluations, blood tests, and an additional sMRI to assess structural changes that may have occurred due to repeated ketamine infusions.

The protocol includes a substudy evaluating ketamine metabolites in healthy volunteers (Ketamine Metabolites Substudy). Only HVs will be enrolled in this substudy. Subjects will undergo a single infusion of ketamine concurrently with serial peripheral blood collection. Some participants may also undergo serial CSF collection during the ketamine infusion. Clinical rating scales, cognitive tasks, MEG, S-EEG, CSF and/or blood draws for pharmacokinetics testing and biomarker analyses will be done.

Outcome Measures

The primary outcome measure of Phase II is the pharmacodynamic fMRI and MEG responses to ketamine compared to placebo. Secondary outcome measures include the difference in Montgomery-Asberg Depression Rating Scale (MADRS) score from baseline to 24 hours between the placebo and ketamine infusion, correlations between an antidepressant response and TMS-EP, S-EEG, neuroimaging, cognitive, and NPU measures. In Phase II, the HVs acts as another level of control to identify a potential neuropharmacodynamic signature associated with an antidepressant response to ketamine.

The primary outcome measure for Phase III is the difference or change in MADRS from baseline to the end of 4 weeks of twice-weekly infusions. Secondary outcome measures include cognitive, TMS-EP, S-EEG, and NPU-threat test measures.

The primary outcome measure for the Ketamine Metabolites Substudy are the levels of ketamine metabolites in CSF and peripheral blood.

Other outcome measures for both Phase II and III include clinical rating scales, neurocognitive tests, ketamine levels, plasma neurochemicals, and peripheral blood biomarkers. Additional outcomes in Phase III are baseline and post-repeated dose infusion MRI scans, and neurocognitive test results. Rating scales are the outcomes measures of Phase IV. Subjects will continue Phase IV for 4 weeks or until relapse (whichever comes first). Additional outcomes for the Ketamine Metabolites Substudy are metabolite levels and clinical rating scales

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion Criteria: All Subjects (Main Study)

1. 18 to 65 years of age.
2. Each subject must have a level of understanding sufficient to agree to all required tests and examinations and sign an informed consent document.
3. All subjects must have undergone a screening assessment under either protocol 01-M-0254, "The Evaluation of Patients with Mood and Anxiety Disorders and Healthy Volunteers" or protocol 17-M-0181 ("Recruitment and Characterization of Research Volunteers for NIMH Intramural Studies").
4. Agree to be hospitalized

Additional Inclusion Criteria: Patients with MDD (Main Study)

1. At the initial study enrollment, subjects must have fulfilled DSM-IV or DSM-5 criteria for Major Depression, single episode or recurrent. Subjects must be experiencing a current major depressive episode of at least 2 weeks duration.
2. At the initial screening and beginning of Phases II and III, subjects must have a baseline score on the MADRS >= 20 and YMRS of < 12.
3. Current or past history of lack of response to one adequate antidepressant trial, operationally defined using the Antidepressant Treatment History Form (ATHF); a failed adequate trial of ECT would count as an adequate antidepressant trial.

Ketamine Metabolites Substudy Inclusion Criteria: Healthy Volunteers

1. 18 to 65 years of age.
2. Each subject must have a level of understanding sufficient to agree to all required tests and examinations and sign an informed consent document.
3. All subjects must have undergone a screening assessment under either protocol 01-M-0254 "The Evaluation of Patients with Mood and Anxiety Disorders and Healthy Volunteers") or 17-M-0181 ("Recruitment and Characterization of Research Volunteers for NIMH Intramural Studies").
4. Agree to be hospitalized.

EXCLUSION CRITERIA:

Additional Exclusion Criteria: Patients with MDD (Main Study)

1. Current diagnosis of Bipolar Disorder including Bipolar I, Bipolar II, or Bipolar NOS diagnoses.
2. Current psychotic features or a diagnosis of Schizophrenia or any other psychotic disorder as defined in the DSM-IV or DSM-5.
3. Subjects with a history of DSM-IV or DSM-5 drug or alcohol dependency or abuse (except for caffeine or nicotine dependence) within the preceding 3 months. In addition, subjects who currently are using drugs (except for caffeine or nicotine) must not have used illicit substances or known drugs of abuse in the 2 weeks prior to screen and must have a negative alcohol and drug urine test (except for prescribed benzodiazepines or stimulants) urine test at screening.
4. Treatment with a reversible MAOI within two weeks prior to Phase II.
5. Subjects who, in the investigator s judgment, pose a current serious suicidal or homicidal risk.

Exclusion Criteria: All Subjects (Main Study)

1. Pregnant or nursing women or women who plan to become pregnant. Women who are able to get pregnant must be willing to use at least one form of effective birth control during the entire period of study participation (or until last clinical labs and rating) and have a negative pregnancy test that was obtained no more than 24 hours prior to MRI and infusion of ketamine.
2. Serious, unstable illnesses including hepatic, renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease, coronary artery disease, atherosclerotic ischemic stroke, and atrial fibrillation), endocrinologic, neurologic, immunologic, or hematologic disease.
3. Clinically significant abnormal laboratory tests.
4. Subjects with one or more seizures without a clear and resolved etiology or current use of medication known to lower seizure threshold. History of seizure (regardless of age or etiology), history of epilepsy in self or first-degree relatives, stroke, brain surgery, head injury, or known structural brain lesion will be excluded from the TMS procedures.
5. Treatment with any other concomitant medication 14 days prior to Phase II. An exception of this would be necessary for those who are taking Fluoxetine or Aripiprazole. Prior to Phase II, treatment with Fluoxetine must be discontinued for at least 5 weeks and treatment with Aripiprazole must be discontinued for at least 3 weeks.
6. Any use of opioid medication in the past 3 months
7. Presence of metallic (ferromagnetic) implants (e.g, heart pacemaker, aneurysm clip) (for subjects doing imaging component of the study only).
8. Presence of any medical illness likely to alter brain morphology and/or physiology (e.g., hypertension, diabetes) even if controlled by medications.
9. Subjects who have hearing loss that has been clinically evaluated and diagnosed
10. Participants who are uncomfortable in small closed spaces (have claustrophobia), unable to lie comfortably supine for up to 90 minutes, and would feel uncomfortable in the MRI machine (for subjects doing imaging component of the study only).
11. Positive HIV test
12. Weight > 119 kg
13. [for participants undergoing NPU Threat Test with Auditory Startle] Known history of hearing loss

Additional Exclusion Criteria: Healthy Volunteers (Main Study)

1. Current or past history of any DSM-IV or DSM-5 Axis I disorder based on clinical assessment and confirmed by a structured diagnostic interview (SCID).

Ketamine Metabolites Substudy Exclusion Criteria: Healthy Volunteers

1. Current or past history of any DSM-IV or DSM-5 Axis I disorder based on clinical assessment and confirmed by a structured diagnostic interview (SCID).
2. Current (within the past 3 months) or past alcohol or substance abuse or dependence diagnosis (except for nicotine or caffeine)
3. Pregnant or nursing women or women who plan to become pregnant. Women who are able to get pregnant must be willing to use at least one form of effective birth control during the 4-days of the study participation (or until last clinical labs and rating) and have a negative pregnancy test that was obtained no more than 24 hours prior to infusion of ketamine.
4. Serious, unstable illnesses including hepatic, renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease, coronary artery disease, atherosclerotic ischemic stroke, and atrial fibrillation), endocrinologic, neurologic, immunologic, or hematologic disease.
5. Clinically significant abnormal laboratory tests.
6. Subjects with one or more seizures without a clear and resolved etiology or current use of medication known to lower seizure threshold.
7. Treatment with any other concomitant medication.
8. Any use of opioid medication in the past 3 months
9. Positive HIV test
10. Weight > 119 kg
11. Presence of metallic (ferromagnetic) implants (e.g, heart pacemaker, aneurysm clip) (for subjects doing neuroimaging component of the study only).
12. Participants who are uncomfortable in small closed spaces (have claustrophobia), unable to lie comfortably supine for up to 90 minutes, and would feel uncomfortable in the MRI machine (for subjects requiring clinical MRI scans for safety and/or structural MRI scans for MEG coregistration).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-05-25 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
To demonstrate more robust neuropharmacodynamic effects measured by neuropharmacodynamic imaging (fMRI+EEG and MEG) of ketamine 0.5 mg/kg as compared to placebo administered over 40 minutes. | Multiple
  Magnetoencephalography (MEG) data
Ketamine Metabolites Substudy: To determine if ketamine metabolites cross the blood brain barrier and enter the brain during ketamine IV administration. | Multiple
  Data from peripheral blood and CSF (in some participants)

SECONDARY OUTCOMES:
To profile ketamine s opioid action based on the PLR using video pupillometry. | Multiple
  Pupil diameter, amplitude of constriction, and constriction velocity
To identify baseline peripheral measures associated with response to the administration of ketamine 0.5 mg/kg, as potential biomarkers of acute (24 hour) treatment response. | Baseline to 24-hours post-ketamine infusion
  Plasma/serum biomarkers
To determine if increases in synaptic plasticity, using electrophysiological measures in response to TMS and in association with sleep (i.e. slow wave sleep EEG activity) are associated with better antidepressant response to 0.5 mg/kg ketamine. | Multiple
  Transcranial Magnetic Stimulation (TMS) and Polysomnography (PSG)/Electroencephalography (EEG) data
Ketamine Metabolites Substudy: To correlate metabolite levels in periphery and CSF with changes in clinical rating scales. | Multiple
  CSF and peripheral blood data, clinical rating scale of depression
To demonstrate enhanced efficacy, as measured by the MADRS, of IV ketamine 0.5 mg/kg in participants with MDD using a psychophysiological technique (i.e. NPU-threat test). | Multiple
  Clinical rating scale of depression

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Zarate, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Clinical and demographic and biomarker participant data collected during the trial, after deidentification
Supporting Information: SAP
Time Frame: Starting within 1 year of completion of the study
Access Criteria: The Branch Chief will review requests and obtain approval by the NIMH/DIRP offices of the Scientific and Clinical Directors and/or the NIH IRB.

REFERENCES:
- [Derived] Moaddel R, Zanos P, Farmer CA, Kadriu B, Morris PJ, Lovett J, Acevedo-Diaz EE, Cavanaugh GW, Yuan P, Yavi M, Thomas CJ, Park LT, Ferrucci L, Gould TD, Zarate CA Jr. Comparative metabolomic analysis in plasma and cerebrospinal fluid of humans and in plasma and brain of mice following antidepressant-dose ketamine administration. Transl Psychiatry. 2022 May 2;12(1):179. doi: 10.1038/s41398-022-01941-x. PMID 35501309
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2017-M-0060.html